CLINICAL TRIAL: NCT03395314
Title: A Randomized Active Placebo Controlled Trial of Ketamine in Borderline Personality Disorder
Brief Title: Ketamine in Borderline Personality Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: assessment of project in wake of covid-19 related interruptions
Sponsor: Yale University (Other)
Collaborators: Nathan Kline Institute for Psychiatric Research (Other); American Foundation for Suicide Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000021457
Record Dates: First submitted 2017-12-22; First posted 2018-01-10 (Actual); Results first posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-05

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline Personality Disorder; Ketamine; Suicide; Social Cognition
MeSH Terms: conditions — Borderline Personality Disorder; Suicide | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- midazolam (Placebo Comparator): Midazolam IV; 0.04mg/kg over 40 minutes
  Interventions: Drug: Midazolam
- low dose ketamine (Active Comparator): ketamine IV; 0.5 mg/kg over 40 minutes
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — 1 single dose of IV ketamine
  Arms: low dose ketamine
Drug: Midazolam — 1 single dose of IV midazolam
  Arms: midazolam

SUMMARY:
The purpose of this study is to test the potential of the rapid-acting anti-depressant ketamine to decrease suicidality in Borderline Personality Disorder (BPD).

The rate of completed suicide in BPD is similar to that of depression or schizophrenia. There is currently no specific medication treatment for BPD.

Ketamine is an FDA-approved anesthetic agent that has been shown to rapidly decrease suicidality and improve mood in people with Major Depressive Disorder (MDD). Though symptoms overlap, effective treatments for MDD and BPD differ. This clinical trial tests if ketamine also decreases suicidality and improves mood in BPD.

This trial will also measure several other outcomes after ketamine versus placebo in BPD: adverse events, BPD symptoms, pain, social cognition, and neuroplasticity.

DETAILED DESCRIPTION:
This clinical trial primarily tests the impact of ketamine on suicidal thoughts in Borderline Personality Disorder (BPD). It also tests the impact of ketamine on symptom intensity (for mood, BPD, and pain symptoms), social cognition, and neuroplasticity in people with BPD.

Suicidal ideation and action are too common in BPD, occurring at rates similar to those in people with depression or schizophrenia. Intensive psychotherapy helps, but many people with BPD do not have access to that treatment, and not everyone responds to psychotherapy if they do get access. No medication is FDA-approved for BPD, and no medication has been shown to decrease suicidality in BPD.

Ketamine is a promising medication for this problem. It is an FDA-approved anesthetic medication with N-methyl D-aspartate activity. Sub-anesthetic doses of ketamine decrease suicidality and improve mood in people with Major Depressive Disorder (MDD). This effect is rapid, with symptom improvement within hours that endures approximately two weeks. People with BPD can have symptoms that overlap with those of MDD, however, the effective treatments for BPD and MDD differ. This clinical trial will test if ketamine, which is effective in MDD, is also effective in BPD.

The investigators will use semi-structured interviews and self-report questionnaires to measure suicidal ideation and clinical symptoms (adverse events, mood symptoms, BPD symptoms, and pain). Social cognition will be also be measured using both interviews/questionnaires and cognitive psychology tasks.

One proposed mechanism of ketamine's effect in MDD is increased neuroplasticity - opening a window during which new learning can occur. This mechanism has been demonstrated in rodent models of depression. In BPD, negatively-biased social interpretations impede meaningful recovery and increase suicide risk over time. A post-ketamine neuro-plastic window may provide an opportunity for revisions of rigid social attributions. The investigators will test for changes in neuroplasticity using a cognitive psychology task and electro-encephalography.

Baseline measures of demographics, life experiences, and symptoms may also be used to predict outcomes or as co-variates in our analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-60
* Clinical diagnosis of Borderline Personality Disorder
* Has suicidal ideation.
* Fluent in English
* Has a current mental health treater, and agrees for study to communicate with treater

Exclusion Criteria:

* Current suicidal intent
* Med changes in last 4 weeks
* Any ketamine in any context in the last one year.
* Current prescription for topiramate, lamotrigine, or lithium.
* Psychotic disorder in self or first-degree relative
* Current substance dependence including alcohol dependence
* Any history of NMDA (N-methyl-D-aspartate )-antagonist abuse
* Any history of opiate abuse
* History of major medical illness especially neurologic or cardiovascular condition, or any other medical contra-indication to ketamine administration at the discretion of the study MD.
* Positive urine test for drugs of abuse screening on day of ketamine administration
* Positive pregnancy test on day of ketamine administration
* At the discretion of study staff

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Fineberg, MD/PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Connecticut Mental Health Center, New Haven, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Midazolam | Low Dose Ketamine
Started | 12 | 10
Completed | 12 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Midazolam | Low Dose Ketamine | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (11.4) | 32.1 (10.4) | 33.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  Arabic | 0 | 1 | 1
  White | 10 | 9 | 19
  Hispanic | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 10 | 22
Education (years) [Mean (Standard Deviation); unit: years] | 16.3 (2.7) | 15.0 (2.7) | 15.7 (2.7)
Baseline Comorbidities [Count of Participants; unit: Participants]
  Major Depressive Disorder | 5 | 5 | 10
  Post-Traumatic Stress Disorder | 4 | 3 | 7
  Anxiety Disorders | 9 | 7 | 16
  Mild Substance Use Disorder | 3 | 3 | 6
  Bipolar Disorder | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Suicidal Thoughts as Measured by Item 10 on the Montgomery-Asberg Depression Scale (MADRS)
Description: The MADRS test includes 10 items and uses a 0 to 6 severity scale for each item, with higher scores indicating increasing depressive symptoms. Scores are averaged across items and can range from 0 to 6 (with 0 indicating enjoying life, and 6 indicating explicit plans for suicide). Outcome description updated when results were entered.
Time Frame: Timepoints will be baseline, 1hr post-infusion and at 1, 3, 7, 14, & 28 days after infusion.
Population: Intention to treat.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Midazolam | Low Dose Ketamine
Number analyzed (Participants) | 12 | 10
units on a scale
  baseline | 2.66 (0.37) | 2.7 (0.41)
  1hr post-infusion | 0.0 (0.37) | 0.1 (0.41)
  Day 1 post-infusion | 0.59 (0.38) | 0.5 (0.41)
  Day 3 post-infusion | 0.89 (0.38) | 0.7 (0.41)
  Day 7 post-infusion | 0.83 (0.37) | 0.8 (0.41)
  Day 14 post-infusion | 1.66 (0.37) | 1.3 (0.41)
  Day 28 post-infusion | 1.29 (0.4) | 2.6 (0.42)

2. Primary Outcome: Change in Suicidality as Measured by the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: Suicide Rating Scale from 1-5; higher numbers indicate increased suicidal thinking.
Time Frame: Timepoints will be baseline, 1hr post-infusion and at 1, 3, 7, 14, & 28 days after infusion.
Population: Intention to treat.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Midazolam | Low Dose Ketamine
Number analyzed (Participants) | 12 | 10
score on a scale
  baseline | 1.58 (0.31) | 1.9 (0.34)
  1hr post-infusion | 0 (0.31) | 0.0 (0.34)
  Day 1 post-infusion | 0 (0.31) | 0.0 (0.34)
  Day 3 post-infusion | 0.75 (0.31) | 0.5 (0.34)
  Day 7 post-infusion | 0.83 (0.31) | 0.3 (0.34)
  Day 14 post-infusion | 0.91 (0.31) | 0.8 (0.34)
  Day 28 post-infusion | 1.16 (0.31) | 1.6 (0.34)

3. Primary Outcome: Change in Suicidality as Measured by Item-12 on the Quick Inventory of Depressive Symptomatology (QIDS SR-16)
Description: The Quick Inventory of Depressive Symptomatology (QIDS SR-16) is a a self-report measure of depression. Each item is scored from 0-3. Higher scores denote more severe load of depressive symptoms. Item 12 measures thoughts of death or suicide from 0 (no thoughts) to 3 (specific suicide plan or action.). Presented is the mean score across items with a range of 0 to 3 where the higher score indicates greater depressive symptoms. Outcome description was updated at the time of results entry.
Time Frame: Timepoints will be baseline, 1hr post-infusion and at 1, 3, 7, 14, & 28 days after infusion.
Population: Intention to treat.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Midazolam | Low Dose Ketamine
Number analyzed (Participants) | 12 | 10
score on a scale
  baseline | 1.25 (0.21) | 1.5 (0.23)
  1hr post-infusion | 0.08 (0.21) | 0.2 (0.23)
  Day 1 post-infusion | 0.34 (0.21) | 0.1 (0.23)
  Day 3 post-infusion | 0.33 (0.21) | 0.3 (0.23)
  Day 7 post-infusion | 0.34 (0.21) | 0.5 (0.23)
  Day 14 post-infusion | 0.71 (0.21) | 0.7 (0.23)
  Day 28 post-infusion | 0.55 (0.22) | 1.21 (0.23)

4. Primary Outcome: Change in Suicidality as Measured by Item 9 on Beck Depression Inventory
Description: When the test is scored, a value of 0 to 3 is assigned for each answer and then the total score is used to quantify the participant's degree of depression from 0 = no depression to 63 = maximally severe depression. Item 9 measures degree of suicidal thoughts or wishes from 0 = no thoughts to 3 = suicidal intent.
Time Frame: Timepoints will be baseline, 1hr post-infusion and at 1, 3, 7, 14, & 28 days after infusion.
Population: Intention to treat.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Midazolam | Low Dose Ketamine
Number analyzed (Participants) | 12 | 10
units on a scale
  baseline | 1.16 (0.19) | 1.2 (0.21)
  1hr post-infusion | 0.08 (0.19) | 0.1 (0.21)
  Day 1 post-infusion | 0.36 (0.19) | 0.3 (0.21)
  Day 3 post-infusion | 0.24 (0.19) | 0.3 (0.21)
  Day 7 post-infusion | 0.41 (0.19) | 0.3 (0.21)
  Day 14 post-infusion | 0.5 (0.19) | 0.3 (0.21)
  Day 28 post-infusion | 0.70 (0.19) | 0.56 (0.21)

5. Secondary Outcome: Change in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS scale measures the depression level of a participant. The total score was derived by adding the scores of the following 10 items: 1, Apparent sadness; 2, Reported sadness; 3, Inner tension; 4, Reduced sleep; 5, Reduced appetite; 6, Concentration difficulties; 7, Lassitude; 8, Inability to feel; 9, Pessimistic thoughts; 10, Suicidal thoughts. Each item was scored using a scale of 0 to 6 (a higher score indicates increased severity). The maximum total score is 60; 0, no depression; 60, severely depressed.
Time Frame: Timepoints will be baseline, 1hr post-infusion and at 1, 3, 7, 14, & 28 days after infusion.
Population: Intention to treat.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Midazolam | Low Dose Ketamine
Number analyzed (Participants) | 12 | 10
score on a scale
  Baseline | 26.75 (2.71) | 28.3 (2.97)
  1hr post-infusion | 3.66 (2.71) | 6.2 (2.97)
  Day 1 | 9.27 (2.78) | 8.2 (2.97)
  Day 3 | 11.70 (2.78) | 12.2 (2.97)
  Day 7 | 12.5 (2.71) | 12.3 (2.97)
  Day 14 | 19.25 (2.71) | 12.9 (2.97)
  Day 28 | 17.39 (2.85) | 22.67 (3.06)

6. Secondary Outcome: Change in Beck Depression Inventory Score
Description: The Beck Depression Inventory (BDI) consisted of twenty-one questions about how the subject has been feeling in the last week. Each question has a set of at least four possible answer choices, ranging in intensity.
  When the test is scored, a value of 0 to 3 is assigned for each answer and then the total score is used to quantify the participant's degree of depression from 0 = no depression to 63 = maximally severe depression.
Time Frame: Timepoints will be baseline, 1hr post-infusion and at 1, 3, 7, 14, & 28 days after infusion.
Population: Intention to treat.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Midazolam | Low Dose Ketamine
Number analyzed (Participants) | 12 | 10
score on a scale
  Baseline | 30.75 (3.96) | 34.9 (4.34)
  1hr post-infusion | 11.16 (3.96) | 13.3 (4.34)
  Day 1 | 12.41 (4.04) | 12.2 (4.34)
  Day 3 | 10.94 (4.04) | 8.9 (4.34)
  Day 7 | 11.33 (3.96) | 12.6 (4.34)
  Day 14 | 17.41 (3.96) | 14.5 (4.34)
  Day 28 | 17.57 (4.04) | 18.73 (4.44)

7. Secondary Outcome: Change in Beck Anxiety Inventory Score
Description: The Beck Anxiety Inventory (BDI) consisted of twenty-one questions about how the subject has been feeling in the last week. Each question has a set of at least four possible answer choices, ranging in intensity.
  When the test is scored, a value of 0 to 3 is assigned for each answer and then the total score is used to quantify the participant's degree of anxiety from 0 = no anxiety to 63 = maximally severe anxiety.
Time Frame: Timepoints will be baseline, 1hr post-infusion and at 1, 3, 7, 14, & 28 days after infusion.
Population: Intention to treat.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Midazolam | Low Dose Ketamine
Number analyzed (Participants) | 12 | 10
score on a scale
  Baseline | 21.75 (2.51) | 21.7 (2.75)
  1hr post-infusion | 4.0 (2.51) | 7.3 (2.75)
  Day 1 | 7.43 (2.57) | 8.3 (2.75)
  Day 3 | 5.71 (2.71) | 5.5 (2.75)
  Day 7 | 7.43 (2.57) | 8.2 (2.75)
  Day 14 | 8.88 (2.57) | 11.0 (2.75)
  Day 28 | 6.34 (2.65) | 18.23 (2.91)

8. Secondary Outcome: Change in Zanarini Rating Scale for Borderline Personality Disorder
Description: A dimensional self-report measure of BPD symptoms that consists of 9 items scored on a 4 point likert scale. Scores range of 0 = minimally symptomatic to 28 = maximally symptomatic for symptoms of Borderline Personality Disorder. Originally, 1hr post-infusion was included as a time frame but this was not collected at this time frame.
Time Frame: Timepoints will be baseline and at 1, 3, 7, 14, & 28 days after infusion.
Population: Intention to treat.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Midazolam | Low Dose Ketamine
Number analyzed (Participants) | 12 | 10
score on a scale
  Baseline | 14.33 (1.78) | 15.4 (1.95)
  Day 1 | 3.52 (1.81) | 5.2 (1.95)
  Day 3 | 5.04 (1.81) | 5.2 (1.95)
  Day 7 | 5 (1.78) | 6.8 (1.95)
  Day 14 | 6.75 (1.78) | 7.2 (1.95)
  Day 28 | 7.16 (1.81) | 11.42 (1.99)

9. Secondary Outcome: Change in Preferred Distance in Stop-distance Paradigm (SDP)
Description: The stop-distance paradigm is a measure of preferred interpersonal distance (PID). Subjects begin the task standing face-to-face and 6 feet away from a test confederate. On each of 3 trials, the confederate slowly approaches the subject. The subjects are instructed to say "stop" to indicate their 1) preferred conversational distance, then a closer distance 2) "if you start to feel uncomfortable". After each "stop", toe to toe distance is measured using a tape measure, and mean PID for the three trials is computed separately for conversational and uncomfortable distance. A computerized version of the task may also be implemented for remote visits and administered in place of the in-person task.
Time Frame: Timepoints will be at baseline and 3, 7, 14, 28 days after infusion
Population: Intention to treat.
Measure: Least Squares Mean (Standard Error); unit: distance in inches
Arm/Group | Midazolam | Low Dose Ketamine
Number analyzed (Participants) | 12 | 10
distance in inches
  Baseline | 18.6 (1.97) | 20.6 (2.5)
  Day 3 | 17.3 (2.12) | 17.2 (2.5)
  Day 7 | 14.7 (2.11) | 15.5 (2.5)
  Day 14 | 19.4 (1.97) | 16.5 (2.5)
  Day 28 | 17.2 (2.11) | 19.5 (2.63)

10. Secondary Outcome: Change in Behavior in the Economic Trust Game - Cooperation
Description: The trust game is a multi-round economic exchange game. There are two roles in the game: investor and trustee. Study participants will play as the trustee. Each round, the investor is given a set number of points and can send any amount to the trustee. The investment triples and the trustee decides how much to repay the investor. Outcome measures are cooperation (amount returned to the investor) and coaxing (amount returned to investor on trials when poor prior returns from trustee have led investor to decrease investment). Cooperation was used as part of the evaluation in this study- coaxing was not. Outcome measure description was updated at the time of results entry.
Time Frame: Timepoints will be at baseline and 3, 7, 14, 28 days after infusion
Population: Intention to treat.
Measure: Least Squares Mean (Standard Error); unit: proportion of amount returned
Arm/Group | Midazolam | Low Dose Ketamine
Number analyzed (Participants) | 12 | 10
proportion of amount returned
  Baseline | 0.39 (0.05) | 0.38 (0.06)
  Day 3 | 0.36 (0.05) | 0.42 (0.06)
  Day 7 | 0.42 (0.05) | 0.29 (0.06)
  Day 14 | 0.34 (0.05) | 0.39 (0.06)
  Day 28 | 0.31 (0.09) | 0.31 (0.06)

11. Secondary Outcome: Change in Social Adjustment Scale Self Report (SAS-SR) Short Version Score
Description: This questionaire measures expressive and instrumental performance over the past two weeks in six role areas: (1) work, either as a paid worker, unpaid homemaker, or student, (2) social and leisure activities, (3) relationships with extended family, (4) role as a marital partner, (5) parental role, and (6) role within the family unit, including perceptions about economic functioning.Each question is rated on a five-point scale from which role area means and an overall mean can be obtained, with higher scores denoting greater impairment. Role areas not relevant to the respondent can be skipped. Overall means are based on all items completed by the respondent. Scores range from 0 = no difficulties to 125 = broad difficulties in multiple domains. An overall adjustment
Time Frame: Timepoints will be at baseline and 3, 7, 14, 28 days after infusion
Population: Intention to treat.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Midazolam | Low Dose Ketamine
Number analyzed (Participants) | 12 | 10
score on a scale
  Baseline | 2.86 (0.18) | 2.74 (0.20)
  Day 3 | 2.30 (0.19) | 1.95 (0.20)
  Day 7 | 2.17 (0.19) | 2.02 (0.20)
  Day 14 | 2.58 (0.18) | 2.07 (0.20)
  Day 28 | 2.33 (0.19) | 2.12 (0.20)

12. Secondary Outcome: Change in Brief Pain Inventory Score - Intensity
Description: Self report inventory that assesses intensity of pain and its interference with everyday life.
  Intensity: pain severity as measured by a 0 to 10 visual analogue scale. 0 = no pain, 10 = worst pain imaginable.
  Interference score: Interference as measured by a 0 to 10 numerical rating scale. 0 = does not interfere, 10 = completely interferes
Time Frame: Timepoints will be at baseline, and post-infusion 1hr, and days 1, 3, 7, 14, & 28.
Population: Intention to treat.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Midazolam | Low Dose Ketamine
Number analyzed (Participants) | 12 | 10
score on a scale
  Baseline | 6.19 (0.93) | 6.32 (1.03)
  Post-infusion 1hr | 5.75 (1.64) | 2.56 (2.23)
  Day 1 | 6.52 (1.34) | 4.46 (2.28)
  Day 3 | 6.73 (1.61) | 4.46 (2.28)
  Day 7 | 9.04 (2.22) | 5.92 (1.16)
  Day 14 | 3.2 (1.33) | 4.14 (1.16)
  Day 28 | 6.28 (1.62) | 5.11 (1.33)

13. Secondary Outcome: Change in Brief Pain Inventory Score - Interference
Description: as for outcome 12
Time Frame: Timepoints will be at baseline, and post-infusion 1hr, and days 1, 3, 7, 14, & 28.
Population: Intention to treat.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Midazolam | Low Dose Ketamine
Number analyzed (Participants) | 12 | 10
score on a scale
  Baseline | 3.49 (1.05) | 2.94 (1.13)
  Post-infusion 1hr | 1.22 (1.58) | 0.51 (1.94)
  Day 1 | 4.79 (1.34) | 3.1 (2.03)
  Day 3 | 3.41 (1.51) | 3.1 (2.03)
  Day 7 | 4.06 (1.95) | 4.09 (1.36)
  Day 14 | 2.21 (1.36) | 3.45 (1.19)
  Day 28 | 4.23 (1.64) | 4.52 (1.36)

14. Secondary Outcome: Change in Clinician-Administered Dissociative States Scale (CADSS) Score
Description: This scale captures the range of possible subjective side effects of ketamine or Midazolam. This consists of 23 questions and scores for each question range from 0-4. The maximum score is 92 with higher scores indicating more dissociative symptoms.
Time Frame: Timepoints: pre- infusion, during infusion +20, +40 minutes, and post-infusion 40 minutes.
Population: Intention to treat.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Midazolam | Low Dose Ketamine
Number analyzed (Participants) | 12 | 10
score on a scale
  Baseline (pre-infusion) | 5.94 (4.11) | 5.92 (3.99)
  20 minutes (during infusion) | 5.54 (3.46) | 25.4 (3.63)
  40 minutes (during infusion) | 9.54 (3.46) | 16.8 (3.63)
  80 minutes (post infusion) | 1.90 (3.46) | 3.0 (3.63)

15. Secondary Outcome: Change in Adverse Events
Description: Adverse events were tracked in a log of treatment emergent adverse events, EKG, pulse oximetry, vital signs. A count of any treatment emergent adverse events is presented through Day 28. The outcome measure description as updated when results were entered.
Time Frame: Timepoints: Continuous monitoring throughout infusion; post-infusion days 1, 3, 7, 14, 28.
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam | Low Dose Ketamine
Number analyzed (Participants) | 12 | 10
Participants | 0 | 0

16. Secondary Outcome: Change in 'Reading the Mind in the Eyes' Test (RMET) Score
Description: The RMET is an advanced test of theory of mind. It is widely used to assess individual differences in social cognition and emotion recognition across different groups and cultures. This is a score from 0-36 where higher score indicates better performance.
Time Frame: Timepoints: at baseline and 3, 7, 14, 28 days after infusion.
Population: Intention to treat.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Midazolam | Low Dose Ketamine
Number analyzed (Participants) | 12 | 10
score on a scale
  Baseline | 28.2 (1.11) | 25.6 (1.23)
  Day 3 | 27.6 (1.13) | 27.3 (1.23)
  Day 7 | 29.2 (1.11) | 26.6 (1.23)
  Day 14 | 29.9 (1.11) | 25.1 (1.23)
  Day 28 | 29.9 (1.11) | 25.4 (1.26)

17. Secondary Outcome: Change in Brief Psychiatric Rating Scale (BPRS) Total Scores
Description: BPRS is an 18-item clinician rated scale with 11 general symptom items, 5 positive-symptom items, and 2 negative symptom items scored on a 7-point scale (1=not present and 7=extremely severe), with higher score indicating greater severity of symptom. Total possible score range=18 to 126.
Time Frame: Timepoints: pre-infusion, during infusion +20, +40 minutes, post-infusion +40 minutes
Population: Intention to treat.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Midazolam | Low Dose Ketamine
Number analyzed (Participants) | 12 | 10
score on a scale
  Baseline (pre-infusion) | 29.36 (2.34) | 33.79 (2.20)
  20 Minutes (during infusion) | 28.18 (1.81) | 38.7 (1.90)
  40 Minutes (during infusion) | 28.0 (1.81) | 36.2 (1.90)
  80 Minutes (post infusion) | 25.9 (1.81) | 28.2 (1.90)

18. Secondary Outcome: Change in Beck Suicide Scale Total Score
Description: The Beck Suicide Scale is a 23 item self report scale with items to specifically assess the presence and intensity of thoughts and actions related to suicidality. Each item response is on a 3 point likert (0-2) for each of 21 items, so possible totals range from 0-42. Higher scores indicate higher suicidality. The description was updated when results were entered.
Time Frame: Timepoints will be baseline, 1hr post-infusion and at 1, 3, 7, 14, & 28 days after infusion.
Population: Intention to treat.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Midazolam | Low Dose Ketamine
Number analyzed (Participants) | 12 | 10
score on a scale
  Baseline | 7.66 (1.75) | 11.5 (1.91)
  1hr post-infusion | 3.5 (1.75) | 4.1 (1.91)
  Day 1 | 3.13 (1.79) | 3.3 (1.91)
  Day 3 | 2.92 (1.79) | 3.9 (1.91)
  Day 7 | 3.08 (1.75) | 4.6 (1.91)
  Day 14 | 5.66 (1.75) | 5.4 (1.91)
  Day 28 | 4.51 (1.79) | 7.12 (1.97)

19. Other Pre Specified Outcome: Change in Bias Scores on the Implicit Association Tests (IAT) of Death, Escape and Self Harm Imagery.
Description: The Implicit Association Test measures implicit automatic associations by tracking the speed at which participants associate different groups of words. The scale is delivered electronically using an open-source software. Three distinct IATs will be administered to assess participant's implicit associations with death, escape, and self harm imagery respectively.
Time Frame: Timepoints: at baseline and 1, 3, 7, 28 days after infusion.
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Change in Resting State Electroencephalography (EEG)
Description: measurement of electrical patterns in the brain while subject is at rest with eyes open looking at fixation cross
Time Frame: Timepoints: at baseline and 1 and/or 7 days after infusion.
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Change in Electroencephalography (EEG) Signal During Behavioral Neuroplasticity Task
Description: measurement of electrical patterns in the brain while subject is performing behavioral task to measure basic neuroplasticity
Time Frame: Timepoints: at baseline and 1 and/or 7 days after infusion.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Uo to 28 days
Arm/Group | Midazolam | Low Dose Ketamine
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 7/12 | 6/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Midazolam (N=12) | Low Dose Ketamine (N=10)
Vivid dreams (Nervous system disorders) | 7 (13) | 6 (23)
Blurry/double vision (Nervous system disorders) | 2 (3) | 3 (9)
Jerky muscle movements (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (10)
Nausea or vomiting (Gastrointestinal disorders) | 3 (10) | 4 (12)
Diarrhea (Gastrointestinal disorders) | 2 (6) | 1 (1)
Hallucinations/Misperceptions (Nervous system disorders) | 0 (0) | 1 (1)
Headaches (Nervous system disorders) | 4 (8) | 1 (2)
Fatigue/Unsteadiness (Nervous system disorders) | 4 (6) | 2 (2)
Increased thirst (Endocrine disorders) | 0 (0) | 1 (1)
Body pain (Nervous system disorders) | 0 (0) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT03395314/Prot_SAP_000.pdf